CLINICAL TRIAL: NCT04979377
Title: Prevalence of Hyperandrogenism in Young Women With Type 1 Diabetes and Study of the Underlying Pathophysiological Mechanisms
Brief Title: Prevalence of Hyperandrogenism in Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Collaborators: Hospital Universitario Ramon y Cajal (Other); Spanish Biomedical Research Centre in Diabetes and Associated Metabolic Disorders (Other); University of Alcala (Other); Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Manuel Luque Ramírez, Co-Principal investigator, Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal
Other Study IDs: DM1PCOS
Record Dates: First submitted 2021-07-07; First posted 2021-07-28 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Type 1 Diabetes; Polycystic Ovary Syndrome; Hyperandrogenism; Hirsutism; Oligomenorrhea; Ovulation Disorder
Keywords: Polycystic ovary syndrome; Hyperandrogenism; Type 1 diabetes; Prevalence; Hirsutism; Ovulatory dysfunction; Testosterone; Insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Polycystic Ovary Syndrome; Hyperandrogenism; Hirsutism; Oligomenorrhea; Insulin Resistance | interventions — Body Mass Index; Body Composition; Cardiovascular Physiological Phenomena; Waist Circumference; Waist-Hip Ratio; Time; Insulin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Serum, plasma and DNA archive samples for further analyses. Registry number (Instituto de Salud Carlos III): C.0005860
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adult premenopausal women with type 1 diabetes mellitus: One-hundred and fifty women aged from 18 to 45 years old consecutively recruited from a type 1 diabetes clinic at a tertiary hospital of Madrid, Spain
  Interventions: Other: Clinical hyperandrogenism assessment; Diagnostic Test: Total testosterone (ng/dL); Diagnostic Test: A1c (%); Diagnostic Test: Total cholesterol; Other: Body mass index (BMI) (kg/m2); Diagnostic Test: Frequency of chronic vascular complications [n (%)]; Diagnostic Test: Polycystic ovary morphology; Diagnostic Test: Cardiovascular autonomic reflex tests (CARTs); Diagnostic Test: Sex hormone-binding globulin (SHBG) (nmol/L); Diagnostic Test: Dehydroepiandrosterone-sulphate (IQL) (ng/mL); Other: Waist circumference (cm); Other: Waist-to-hip ratio; Other: Body composition; Diagnostic Test: Mean glucose (mg/dL); Diagnostic Test: Time in target range (hours); Diagnostic Test: Time in hyperglycemia (hours); Other: Insulin dose (UI/Kg); Other: Insulin sensitivity; Diagnostic Test: High-density lipoprotein (HDL) (mg/dL); Diagnostic Test: Low-density lipoprotein (LDL) (mg/dL); Diagnostic Test: Triglycerides (mg/dL)

INTERVENTIONS:
Other: Clinical hyperandrogenism assessment — Modified Ferriman-Gallwey scale
  Other Names: Hirsutism score
Diagnostic Test: Total testosterone (ng/dL) — Circulating total testosterone (LC-MS/MS or IQL-CDC method) at follicular phase
  Other Names: Sex steroid profile
Diagnostic Test: A1c (%) — High Performance Liquid Chromatography (HPLC)
  Other Names: Metabolic control
Diagnostic Test: Total cholesterol — Determined by enzymatic methods
  Other Names: Lipid profile
Other: Body mass index (BMI) (kg/m2) — Defined as body weight divided by the square of body height, and expressed in kg/m2
  Other Names: Anthropometrics and body composition
Diagnostic Test: Frequency of chronic vascular complications [n (%)] — Retinopathy, nephropathy, neuropathy, and macrovascular disease.
Diagnostic Test: Polycystic ovary morphology — Sonographic assessment
Diagnostic Test: Cardiovascular autonomic reflex tests (CARTs) — Cardioautonomic function assessement by Vital scan HW7-HW6T:
  Other Names: Cardiovascular function
Diagnostic Test: Sex hormone-binding globulin (SHBG) (nmol/L) — Circulating SHBG (IQL) at follicular phase
  Other Names: Sex steroid profile
Diagnostic Test: Dehydroepiandrosterone-sulphate (IQL) (ng/mL) — Circulating DHEAS (IQL) at follicular phase
  Other Names: Sex steroid profile
Other: Waist circumference (cm) — Waist circumference measurement made at the top of the iliac crest
  Other Names: Anthropometrics and body composition
Other: Waist-to-hip ratio — Waist circumference divided by hip circumference (measurement should be taken around the widest portion of the buttocks)
  Other Names: Anthropometrics and body composition
Other: Body composition — Vital Scan HW7-HW6T
  Other Names: Bioimpedanciometry
Diagnostic Test: Mean glucose (mg/dL) — Continuous glucose monitoring (GCM) records
  Other Names: Metabolic control
Diagnostic Test: Time in target range (hours) — Continuous glucose monitoring (GCM) records
  Other Names: Metabolic control
Diagnostic Test: Time in hyperglycemia (hours) — Continuous glucose monitoring (GCM) records
  Other Names: Metabolic control
Other: Insulin dose (UI/Kg) — Daily insulin dose divided by body weight
  Other Names: Metabolic control
Other: Insulin sensitivity — Equation that relies on routine clinical measures: A1c, presence of hypertension, and waist circumference
  Other Names: Estimated glucose disposal rate (eGDR)
Diagnostic Test: High-density lipoprotein (HDL) (mg/dL) — Enzymatic methods after precipitation of serum with phosphotungstic acid and Mg2+
  Other Names: HDL-cholesterol
Diagnostic Test: Low-density lipoprotein (LDL) (mg/dL) — Estimated by the Friedewald's equation.
  Other Names: Lipid profile
Diagnostic Test: Triglycerides (mg/dL) — Determined by enzymatic methods
  Other Names: Lipid profile

SUMMARY:
The investigators aim to estimate the prevalence of functional ovarian hyperandrogenism [idiopathic hyperandrogenism, idiopatic hirsutism, and polycystic ovary syndrome (PCOS)] in adult patients with type 1 diabetes (T1DM) in an observational cross-sectional study. Study population is comprised of premenopausal adult women with a diagnosis of T1DM, consecutively recruited from a Diabetes outpatient clinic at a tertiary hospital in Spain, Europe.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is the most common endocrine disorder in women of reproductive age, with an estimated prevalence of 6-15% of the general population worldwide. This heterogeneous syndrome has significant cardio-metabolic, reproductive, and psycho-emotional consequences, and therefore, a prompt recognition and management is of paramount importance for these women. Despite hyperandrogenism is the cornerstone in the pathophysiology of PCOS, this derangement is closely related to insulin resistance, compensatory hyperinsulinemia, and abdominal adiposity. Hyperinsulinemia increases androgen secretion by co-stimulating besides gonadotropins both ovary and adrenal steroidogenesis, which leads to predominant visceral/abdominal fat deposition, and further contributes to insulin resistance and hyperinsulinemia. In addition, PCOS has been classically associated with metabolic alterations such as for overweight/obesity and type 2 diabetes mellitus. However, type 1 diabetes mellitus (T1D) results from autoimmune-mediated destruction of the pancreas, causing a complete insulin lack in most patients. Intensive insulin therapy - a mandatory iatrogenic hyperinsulinism -, while improving chronic glycemic control and prognosis, has led in recent years to the appearance of "new" reproductive consequences in these patients, such as functional hyperandrogenism and menstrual irregularity. This association is expected from the stimulation of ovarian androgen production by exogenous insulin, which reaches the ovary in supraphysiological concentrations. However, these studies present with a high heterogeneity, and prevalence rates significantly vary depending on several variables such as the criteria used for PCOS diagnosis, race/ethnicity, age of the study population, and the prevalence of obesity, among others. In 2016, a systematic review assessing the prevalence of PCOS in T1D was published, including 475 women with T1D from 9 studies. The results showed an overall prevalence of PCOS about 24% in T1D, higher than reported in the general population. Other hyperandrogenic traits such as hirsutism (25%), hyperandrogenaemia (24%), or ovulatory dysfunction (33%) were also common. Although PCOS is one of the most common comorbidities in patients with T1D, there are a limited number of publications in the literature. In summary, PCOS and functional hyperandrogenism remain a condition to be explored thoroughly in these patients.

The investigators hypothesize that the prevalence of functional hyperandrogenism including PCOS in Spanish women with T1D is higher than in women from the general population. Furthermore, signs and symptoms of hyperandrogenism, and hyperandrogenemia may be milder in patients with T1D compared to hyperandrogenic women from the general population. Moreover, the occurrence of PCOS in these women may be influenced by insulin dose, duration of diabetes, and chronic metabolic control.

The main objective of this study is to determine the actual prevalence of PCOS in premenopausal women with T1DM, according to different diagnostic criteria/PCOS phenotypes [classic PCOS (classic NIH criteria), hyperandrogenic PCOS (AES-PCOS criteria), and/or inclusive ESHRE-ASRM/Rotterdam criteria]. As secondary goals, the investigators also aim to describe: i) the hyperandrogenic traits associated with PCOS in women with T1DM; and ii) the metabolic-T1D related parameters in women with or without hyperandrogenism.

Sample size calculation: Sample size analysis used the online sample size and power calculator from the Program of Research in Inflammatory and Cardiovascular Disorders, Institut Municipal d'Investigació Mèdica, Barcelona, Spain (https://www.imim.cat/ofertadeserveis/software-public/granmo/). Considering previous data on prevalence of SOP in adolescents and adult women with T1D according to ESHRE-ASRM/Rotterdam criteria, the investigators concluded that 150 participants would be needed to assume an expected proportion of 40%, with an absolute precision of 5% at both sides of the proportion, and an asymptotic bilateral 95% confidence interval, and with an estimated replacement rate of 10%.

Statistical analysis: Continuous variables will be expressed as mean ± SD with its respective 95% confidence intervals (95%CI). Normality of continuous variables will be checked by the Kolmogorov-Smirnov test, and ensured by applying logarithmic transformations. the investigators will use non-parametric tests to analyse variables that remained skewed even after transformation. The differences in means will be analysed by Student t or Mann-Whitney U tests. Discrete variables will be showed according to their absolute, relative frequency, and 95%CI determined using the Wilson method without continuity correction. The differences between proportions will be estimated using the χ2 or Fisher's exact tests. Correlation analysis will be used to evaluate putative association between continuous variables. Finally, multiple linear an binary logistic regression full and stepwise models (probability for entry ≤0.05, probability for removal ≥0.10) will be performed to ascertain the main determinants of predetermined outcomes. The statistical significance will be set at the P < 0.05 level.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 45 years old
* Type 1 diabetes diagnosed at least 1 year before the inclusion in the study. Diagnosis confirmed by positive autoimmunity (GAD-65 or IA2) and insulin deficiency.
* Treatment with subcutaneus insulin therapy (multiple dose or continuous subcutaneous insulin infusion).
* Menarche at least 2 years before the study.

Exclusion Criteria:

* Honey moon period.
* Altered thyroid hormone or prolactin levels.
* Congenital adrenal hyperplasia.
* Severe chronic disease.
* Oral contraceptive or glucocorticoid therapy in the previous 3 months.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Premenopausal women with T1DM consecutively recruited from a Diabetes outpatient clinic at a tertiary hospital.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2020-03-09 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of PCOS in T1DM | 2020-2022
  Prevalence of PCOS in women with T1DM according to ESHRE-ASRM/Rotterdam criteria
Prevalence of classic PCOS in T1DM | 2020-2022
  Prevalence of PCOS in women with T1DM according to classic NIH criteria
Prevalence of hyperandrogenic PCOS in T1DM | 2020-2022
  Prevalence of PCOS in women with T1DM according to AES-PCOS criteria

SECONDARY OUTCOMES:
Prevalence of related traits in women with T1D | 2020-2022
  Prevalence of related hyperandrogenic traits (idiopatic hirsutism, hyperandrogenemia, oligomenorrhea and isolated polycytic ovarian morphology) in women with T1DM
Influence fo the onset of type 1 diabetes on hyperandrogenism | 2020-2022
  To assess the influence of the timing of diagnosis of type 1 diabetes in the appearance of hyperandrogenism, and also the possible effect of duration of diabetes.
Influence of Insulin Requirements on hyperandrogenism | 2020-2022
  To describe daily insulin requirements and their influence on functional hyperandrogenism occurrence. We also aim to determine the effect of the chronic metabolic control in PCOS appearance.
Influence of metabolic control on hyperandrogenism | 2020-2022
  To describe the influence of metabolic control (A1c) on functional hyperandrogenism occurrence. We also aim to determine the effect of the chronic metabolic control in PCOS appearance.
Influence of body composition on hyperandrogenism | 2020-2022
  To evaluate the influence of risk factors body composition in the occurrence of ovarian hyperandrogenism and PCOS in women with type 1 diabetes.
Influence of hyperandrogenism on insulin requirements | 2020-2022
  To describe the influence of hyperandrogenism on metabolic control.
Influence of hyperandrogenism on A1c | 2020-2022
  To describe the influence of hyperandrogenism on metabolic control.
Influence of hyperandrogenism on mean glucose (GCM) | 2020-2022
  To describe the influence of hyperandrogenism on metabolic control.
Influence of hyperandrogenism on time in range (GCM) | 2020-2022
  To describe the influence of hyperandrogenism on metabolic control.
Influence of hyperandrogenism on chronic complications | 2020-2022
  To describe the influence of hyperandrogenism on the frequency of chronic complications related to type 1 diabetes mellitus

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Luque-Ramírez, PhD, MD, MBA, Study Director — CIBERDEM, Instituto de Salud Carlos III; Héctor F Escobar-Morreale, PhD, MD, Study Chair — University of Alcalá
Locations (1):
- Hospital Universitario Ramón y Cajal, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
All data sets generated during and/or analyzed during the current study are not publicly available but are available from the corresponding author on reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Since study ending with no time limit restriction
Access Criteria: Reasonable request

REFERENCES:
- [Background] Escobar-Morreale HF, Roldan B, Barrio R, Alonso M, Sancho J, de la Calle H, Garcia-Robles R. High prevalence of the polycystic ovary syndrome and hirsutism in women with type 1 diabetes mellitus. J Clin Endocrinol Metab. 2000 Nov;85(11):4182-7. doi: 10.1210/jcem.85.11.6931. PMID 11095451
- [Background] Roldan B, Escobar-Morreale HF, Barrio R, de La Calle H, Alonso M, Garcia-Robles R, Sancho J. Identification of the source of androgen excess in hyperandrogenic type 1 diabetic patients. Diabetes Care. 2001 Jul;24(7):1297-9. doi: 10.2337/diacare.24.7.1297. No abstract available. PMID 11423519
- [Background] Codner E, Escobar-Morreale HF. Clinical review: Hyperandrogenism and polycystic ovary syndrome in women with type 1 diabetes mellitus. J Clin Endocrinol Metab. 2007 Apr;92(4):1209-16. doi: 10.1210/jc.2006-2641. Epub 2007 Feb 6. PMID 17284617
- [Background] Escobar-Morreale HF, Roldan-Martin MB. Type 1 Diabetes and Polycystic Ovary Syndrome: Systematic Review and Meta-analysis. Diabetes Care. 2016 Apr;39(4):639-48. doi: 10.2337/dc15-2577. PMID 27208367
- [Background] Codner E, Soto N, Lopez P, Trejo L, Avila A, Eyzaguirre FC, Iniguez G, Cassorla F. Diagnostic criteria for polycystic ovary syndrome and ovarian morphology in women with type 1 diabetes mellitus. J Clin Endocrinol Metab. 2006 Jun;91(6):2250-6. doi: 10.1210/jc.2006-0108. Epub 2006 Mar 28. PMID 16569737
- [Background] Codner E, Iniguez G, Villarroel C, Lopez P, Soto N, Sir-Petermann T, Cassorla F, Rey RA. Hormonal profile in women with polycystic ovarian syndrome with or without type 1 diabetes mellitus. J Clin Endocrinol Metab. 2007 Dec;92(12):4742-6. doi: 10.1210/jc.2007-1252. Epub 2007 Sep 25. PMID 17895317
- [Background] Gaete X, Vivanco M, Eyzaguirre FC, Lopez P, Rhumie HK, Unanue N, Codner E. Menstrual cycle irregularities and their relationship with HbA1c and insulin dose in adolescents with type 1 diabetes mellitus. Fertil Steril. 2010 Oct;94(5):1822-6. doi: 10.1016/j.fertnstert.2009.08.039. Epub 2009 Sep 30. PMID 19796762
- [Background] Codner E, Merino PM, Tena-Sempere M. Female reproduction and type 1 diabetes: from mechanisms to clinical findings. Hum Reprod Update. 2012 Sep-Oct;18(5):568-85. doi: 10.1093/humupd/dms024. Epub 2012 Jun 17. PMID 22709979
- [Background] Nattero-Chavez L, Alonso Diaz S, Jimenez-Mendiguchia L, Garcia-Cano A, Fernandez-Duran E, Dorado Avendano B, Escobar-Morreale HF, Luque-Ramirez M. Sexual Dimorphism and Sex Steroids Influence Cardiovascular Autonomic Neuropathy in Patients With Type 1 Diabetes. Diabetes Care. 2019 Nov;42(11):e175-e178. doi: 10.2337/dc19-1375. Epub 2019 Sep 17. No abstract available. PMID 31530659
- [Background] Teede HJ, Misso ML, Costello MF, Dokras A, Laven J, Moran L, Piltonen T, Norman RJ; International PCOS Network. Recommendations from the international evidence-based guideline for the assessment and management of polycystic ovary syndrome. Hum Reprod. 2018 Sep 1;33(9):1602-1618. doi: 10.1093/humrep/dey256. PMID 30052961
- [Background] Escobar-Morreale HF, Carmina E, Dewailly D, Gambineri A, Kelestimur F, Moghetti P, Pugeat M, Qiao J, Wijeyaratne CN, Witchel SF, Norman RJ. Epidemiology, diagnosis and management of hirsutism: a consensus statement by the Androgen Excess and Polycystic Ovary Syndrome Society. Hum Reprod Update. 2012 Mar-Apr;18(2):146-70. doi: 10.1093/humupd/dmr042. Epub 2011 Nov 6. PMID 22064667
- [Background] Escobar-Morreale HF, Bayona A, Nattero-Chavez L, Luque-Ramirez M. Type 1 diabetes mellitus and polycystic ovary syndrome. Nat Rev Endocrinol. 2021 Dec;17(12):701-702. doi: 10.1038/s41574-021-00576-0. No abstract available. PMID 34561669